CLINICAL TRIAL: NCT07005882
Title: Hormonal Receptor (HR)-Positive HER2 Negative Breast Cancer Patients Treated With Preoperative ELacestrant and PULSAR Adaptive Radiotherapy: a Phase II Study (HELP Trial)
Brief Title: Hormonal Receptor (HR)-Positive HER2 Negative Breast Cancer Patients Treated With Preoperative ELacestrant and PULSAR Radiotherapy
Acronym: HELP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Full Professor, Azienda Ospedaliero-Universitaria Careggi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HELP Trial; 2025-520762-22-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-25; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer Patients; Breast Cancer Early Stage Breast Cancer (Stage 1-3); HR+/HER2- Breast Cancer; Radiation Therapy
MeSH Terms: interventions — elacestrant; DEAE-Dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Preoperative Elacestrant+PULSAR (Experimental)
  Interventions: Drug: Elacestrant; Radiation: PULSAR

INTERVENTIONS:
Drug: Elacestrant — Preoperative treatment
Radiation: PULSAR — Preoperative treatment

SUMMARY:
This is a proof-of-concept phase II trial to assess the safety (as primary endpoint) and clinical efficacy of neoadjuvant therapy with Elacestrant and PULSAR.

The study will enroll 21 postmenopausal patients with early HR+ HER2- node positive BC, clinically staged II-III. Patients will receive Elacestrant 345 mg orally once daily for 24 weeks and PULSAR on the MRI-based breast gross tumor volume (GTVt), consisting of 10 Gy "pulse" every 4 weeks for a maximum of 5 or less in case of radiologic complete response.

Surgery will be planned 24 weeks after Elacestrant initiation and at least 2 weeks from the last pulse and will be performed as per recommended clinical practice. Patients will then receive adjuvant systemic therapy as per standard of care and postoperative RT to the locoregional lymph nodes in case of nodal residual disease, if indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven HR-positive, HER2-negative BC
2. Clinical disease stage II-III
3. Post-menopausal female patients or male patients
4. Eligible for neoadjuvant treatment and subsequent surgery
5. No contraindication to MRI
6. Patient able to understand and follow instructions during the trial
7. Patient able and willing to give written informed consent, signed and dated
8. Patient aged at least 50 years old
9. Patient with tumor accessible for biopsy and surgery
10. Patient with adequate bone marrow function at Screening, confirmed at Baseline, including:

    1. ANC ≥ 1.5 × 109/L; patients with documented benign cyclical neutropenia are eligible if white blood cell count is ≥ 1.5 × 109/L, with ANC ≥ 1.0 × 109/L, leukocytes ≥ 4.0 × 109/L, and lymphocytes ≥ 0.6 × 109/L;
    2. platelets ≥ 100 × 109/L;
    3. hemoglobin ≥ 9 g/dL (may have been transfused);
11. International Normalized Ratio (INR) < 1.5×Upper Limit of Normal (ULN); patients treated with vitamin K antagonist are eligible if INR < 3
12. Patient with adequate hepatic function at Screening, confirmed at Baseline, defined by:

    a. total bilirubin level ≤1.5×ULN; patients with documented Gilbert disease are allowed if total bilirubin ≤3×ULN; aspartate aminotransferase (AST) level ≤2.5×ULN, and alanine aminotransferase (ALT) level ≤2.5×ULN,
13. Patient with adequate renal function at Screening, confirmed at Baseline, defined by eGFR ≥ 30 mL/min using 2021 CKD-EPI creatinine equation
14. Patient with Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
15. Life expectancy of at least 12 months according to the Investigator's judgement

Exclusion Criteria:

* 1. Patients with stage IV disease 2. Patients with a history of any disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, based on the Investigator's judgement, provides a reasonable suspicion of a disease or condition that contraindicates the use of RT and/or Elacestrant or that might affect the interpretation of the trial results or render the patient at high risk for treatment complications.

  3. Patients with any significant co-morbidity which, according to the Investigator's judgement, makes patient compliance to trial conditions unlikely.

  4. Patients with previous malignant disease (other than the tumor disease for this trial) within the last five (5) years (except adequately treated non-melanoma skin cancers and carcinoma in situ of skin, bladder, cervix, colon/rectum, breast, or prostate) unless a complete remission without further recurrence was achieved at least two (2) years prior to Screening, and the patient is deemed to have been cured with no additional therapy required or anticipated to be required.

  5. Patients with a history of uncontrolled intercurrent illness. 6. Patients with a known prior hypersensitivity or contraindications to Elacestrant or any component in its formulations.

  7. Patients with severe acute or chronic medical conditions, including:
  1. Immune colitis
  2. Inflammatory bowel disease
  3. History of severe vomiting or diarrhea not having resolved to Grade 1 at Baseline
  4. Immune pneumonitis
  5. Pulmonary fibrosis
  6. Psychiatric conditions including recent (within the last year) or active suicidal ideation or behavior
  7. Laboratory abnormalities that may increase the risk associated with trial participation or trial treatment administration or may interfere with the interpretation of trial results and, in the judgement of the Investigator, would make the patient inappropriate for entry into this trial.

     8. Patients with a history of small intestine resection surgery or other major gastrointestinal surgery.

     9. Patients with an active infection requiring systemic therapy with antibiotics (at both Screening and Baseline).

     10. Patients with a known history of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome or multi-drug-resistant gram-negative bacteria.

     11. Patients with hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at Screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody Screening test positive).

     12. Patients with increased anesthesiological risk (e.g. known or predicted difficult airway) if general anesthetic is required.

     13. Premenopausal patients (defined as any woman who is not surgically sterile with a hysterectomy and/or bilateral oophorectomy or >12 months of amenorrhea and at least 50 years of age) 14. Patients aged less than 50 years old. 15. Patients with a known history of drug/substance abuse. 16. Patients participating in any other clinical trial within 30 days before Screening.

     17. Patients receiving any other treatment that, in the opinion of the Investigator, might interfere with the trial.

     18. Concomitant use of strong or moderate CYP3A4 inhibitors should be avoided and an alternative concomitant medicinal product with no or minimal potential to inhibit CYP3A4 should be considered.

     19. Concomitant use of strong or moderate CYP3A4 inducers should be avoided and an alternative concomitant medicinal product with no or minimal potential to induce CYP3A4 should be considered.

     20. Patients with a current drug or substance abuse. 21. Patients receiving chronic concurrent therapy within two (2) weeks before the trial treatment or expected therapy during the trial treatment period with:

  <!-- -->

  1. Corticosteroids (except systemic corticosteroids up to 10 mg prednisolone or equivalent daily dose).
  2. Immunosuppressive agents.
  3. Antibiotics.
  4. Any other anticancer therapy or concurrent anticancer treatment. 22. Patients who are unable to understand the protocol requirements, instructions and trial-related restrictions, the nature, scope, and possible consequences of the trial.

     23. Patients who are unlikely to comply with the Protocol requirements, instructions and trial-related restrictions, e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the trial.

     24. Patients with legal incapacity or limited legal capacity. 25. Patients with any condition which results in an undue risk for the patient during the trial participation according to the Investigator.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Elacestrant combined with PULSAR radiation therapy in preoperative setting | Baseline, every two weeks in the pre-operative period, 30 days and 3 months after surgery
  Evaluation of reported adverse events (AEs) and serious adverse events (SAEs), according to CTCAE v5.0.
  Evaluation of changes from Baseline during the Treatment and Follow-up periods.
Safety of Elacestrant combined with PULSAR radiation therapy in preoperative setting | Baseline, every two weeks unitl week 4, then every 4 weeks in the pre-operative period, 30 days and 3 months after surgery
  Evaluation of changes from Baseline during the Treatment and Follow-up periods in:
  - laboratory parameters: hematology (Hemoglobin, HMCV, MCH, MCHC, RBC, WBC with differential count, and platelet count); biochemistry (Sodium, potassium, calcium, chloride, glucose (fasting), anorganic phosphate, cholesterol, triglycerides, total protein, uric acid, urea, creatinine, total bilirubin, alkaline phosphatase, ALT, AST, gamma-GT, LDH, CPK, amylase, and lipase); coagulation (PT, INR and activated partial thromboplastin time); and urinalysis (Leukocytes, nitrite, pH, protein, glucose, ketone, urobilinogen, bilirubin, hemoglobin, erythrocytes, specific gravity.).
  These values will be used to assess the patient's health status and the presence of any adverse events that may have arisen after therapy.
Safety of Elacestrant combined with PULSAR radiation therapy in preoperative setting | Baseline, every two weeks in the pre-operative period, 30 days, 3 months, 6 months and 12 months after surgery
  Evaluation of changes from Baseline during the Treatment and Follow-up periods in:
  - physical examinations: (i.e. ECOG PS 0-5).
Safety of Elacestrant combined with PULSAR radiation therapy in preoperative setting | Baseline, every two weeks until week 4 and then every 4 weeks in the pre-operative period, 30 days, 3 months, 6 months and 12 months after surgery
  Evaluation of changes from Baseline during the Treatment and Follow-up periods in:
  - vital signs: temperature in °C
Safety of Elacestrant combined with PULSAR radiation therapy in preoperative setting | Baseline, at the beginning (week 0) and at the end (week 20) of pre-operative treatment.
  Evaluation of changes from Baseline during the Treatment and Follow-up periods in:
  - electrocardiograms: heart rate, PR/PQ interval, QRS interval, QT interval.
Safety of Elacestrant combined with PULSAR radiation therapy in preoperative setting | Baseline, every two weeks until week 4 and then every 4 weeks in the pre-operative period, 30 days, 3 months, 6 months and 12 months after surgery
  Evaluation of changes from Baseline during the Treatment and Follow-up periods in:
  - vital signs: heart rate in beats/min (bpm).
Safety of Elacestrant combined with PULSAR radiation therapy in preoperative setting | Baseline, every two weeks until week 4 and then every 4 weeks in the pre-operative period, 30 days, 3 months, 6 months and 12 months after surgery
  Evaluation of changes from Baseline during the Treatment and Follow-up periods in:
  - vital signs: blood pressure in mmHg.
Safety of Elacestrant combined with PULSAR radiation therapy in preoperative setting | Baseline, every two weeks until week 4 and then every 4 weeks in the pre-operative period, 30 days, 3 months, 6 months and 12 months after surgery
  Evaluation of changes from Baseline during the Treatment and Follow-up periods in:
  - vital signs: respiratory frequency in breaths/min.
Safety of Elacestrant combined with PULSAR radiation therapy in preoperative setting | Baseline, every two weeks until week 4 and then every 4 weeks in the pre-operative period, 30 days, 3 months, 6 months and 12 months after surgery
  Evaluation of changes from Baseline during the Treatment and Follow-up periods in:
  - vital signs: SpO2 in %.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Careggi Radiation Oncology Unit, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided